CLINICAL TRIAL: NCT03049709
Title: Non-invasive Automated Central Blood Pressure Measurements Using Oscillometric Pulse Wave Analysis - Comparison With Non-Invasive Reference Values
Brief Title: Non-invasive Validation of Non-invasive Central Blood Pressure Measurements Using Oscillometric Pulse Wave Analysis
Acronym: MEASURE-cBP2
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: VA_noninvasive
Record Dates: First submitted 2017-02-06; First posted 2017-02-10 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Arterial Hypertension; Healthy Control; Coronary Heart Disease; Diabetes Mellitus
Keywords: central blood pressure; measurement; oscillometric radial pulse wave analysis
MeSH Terms: conditions — Hypertension; Coronary Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- cardiovascular disease: patients with cardiovascular disease, invasive and non-invasive determination of central blood pressure
- healthy controls: healthy controls, invasive and non-invasive determination of central blood pressure

SUMMARY:
There is growing evidence that central blood pressure is a better predictor of hypertensive end-organ damage and cardiovascular outcome than routine brachial readings.

The investigators aimed to evaluate the accuracy of a novel device for the non-invasive determination of central blood pressure based on automated oscillometric radial pulse wave analysis.

ELIGIBILITY:
Inclusion Criteria:

* cardiovascular disease, diabetes mellitus or healthy control

Exclusion Criteria:

* inability to give informed consent
* hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in-patients and healthy controls (students, hospital staff)
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
agreement of systolic central blood pressure measurements | 15 minutes
agreement of diastolic central blood pressure measurements | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jens J Kaden, MD, Principal Investigator — Universitätsmedizin Mannheim; Joachim Saur, MD, Principal Investigator — Universitätsmedizin Mannheim; Urs Benck, MD, Principal Investigator — Universitätsmedizin Mannheim
Locations (1):
- Universitätsmedizin Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No